CLINICAL TRIAL: NCT00119041
Title: Diabetes Telemedicine Consultation: A Systems Improvement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 03-254
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus Type 2; Diabetes Mellitus, Type 1; Primary Care Provider
Keywords: Diabetes Mellitus; Telemedicine; Referral; Consultation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemedicine CBOC (Experimental): Designated CBOC's were involved in the intervention phase where their Diabetes Mellitus (DM) patients were asked to participate in a telemedicine visit.
  The Behavioral: The Diabetes Treatment Satisfaction Questionnaire given during this phase along with the Behavioral: Diabetes Empowerment Scale and the Behavioral: CBOC's undergo half-day joint-clinics via teleconference.
  Interventions: Behavioral: The Diabetes Treatment Satisfaction Questionnaire; Behavioral: Diabetes Empowerment Scale; Behavioral: CBOC's undergo half-day joint-clinics via teleconference
- Control CBOC (No Intervention): The CBOC's not involved in the intervention phase had their patients not be involved in the telemedicine visit, but traditional education.
- Provider Interviews (No Intervention): Qualitative interviews with providers

INTERVENTIONS:
Behavioral: The Diabetes Treatment Satisfaction Questionnaire — A six question likert scale questionnaire regarding the patients treatment satisfaction. The responses range from very dissatisfied to very satisfied.
  Arms: Telemedicine CBOC
Behavioral: Diabetes Empowerment Scale — A twenty-eight question likert scale questionnaire regarding the patients attitude towards diabetes. The responses range from strongly agree to strongly disagree.
  Arms: Telemedicine CBOC
Behavioral: CBOC's undergo half-day joint-clinics via teleconference — A patient has Diabetes/Endo clinic visit via teleconferencing. A patient is at a CBOC and the Diabetes/Endo physician is at Wade Park.
  Arms: Telemedicine CBOC

SUMMARY:
This study seeks to evaluate and document the processes of outreach consultation through joint-clinics via teleconferencing as an intervention for system improvement in care delivery and management of diabetes mellitus (DM) at a Community Based Outpatient Center (CBOCs).

DETAILED DESCRIPTION:
Background:

Diabetes is a national problem that has reached epidemic proportions, according to the U.S. Centers for Disease Control and Prevention. Diabetes has particular importance for the Department of Veterans Affairs (VA) because the prevalence among VA patients -- one in six, or 16 percent -- is substantially higher than in the general population.

Objectives:

The objective of this study was to evaluate and document the processes of outreach consultation through the use of joint-clinics via teleconferencing as an intervention for system improvement in care delivery and management of diabetes at CBOCs. The intervention consisted of a teleconferenced joint-clinic consultation session involving the patient, Diabetes Specialist Team, the Primary Care Provider (PCP) and other relevant care team members. The impact of the 16-month intervention was assessed based on patients who were involved in the telemedicine clinic and those who were referred to a specialist to be seen on-site at the Cleveland VAMC.

Methods:

Study settings include the CBOCs affiliated with the Cleveland Veterans Affairs Medical Center (VAMC) and involve primary care referrals to see diabetes specialists at the Cleveland VAMC. Inclusion criteria patients(N 282)=included: (i) current prescription of insulin or an oral hypoglycemic agent; (ii) A1c > 7.0%; or (iii) fasting glucose levels> 130 mg/dl; and (iv) referred to see a consultant (beginning three months prior to the active intervention phase and continuing through enrollment for the last month of the active intervention phase). Patients with either Type l or Type II diabetes will be included. Patients referred will be contacted and asked to participate.

ELIGIBILITY:
Inclusion Criteria:

* 1) Current prescription of insulin or an oral hypoglycemic agent
* 2) A1c > 7.0%
* 3) fasting glucose levels > 130 mg/dl
* 4) referred to see a consultant and are seen during the active intervention phase. Patients with either Type I or Type II DM will be included

A Primary Care Provider for a Cleveland CBOC

Exclusion Criteria:

* 1) primary care obtained at more than one site (based on stop codes with evidence of more than 1 CBOC involved in care during the last 6 months)
* 2) documented dementia, aphasia, and psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Aron, MD MS, Principal Investigator — Louis Stokes VA Medical Center
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Louis Stokes VA Medical Center, Cleveland, Ohio

REFERENCES:
- [Result] Tomolo AM, Lawrence RH, Aron DC. A case study of translating ACGME practice-based learning and improvement requirements into reality: systems quality improvement projects as the key component to a comprehensive curriculum. Qual Saf Health Care. 2009 Jun;18(3):217-24. doi: 10.1136/qshc.2007.024729. PMID 19468006
- [Result] Pogach L, Aron D. Balancing hypoglycemia and glycemic control: a public health approach for insulin safety. JAMA. 2010 May 26;303(20):2076-7. doi: 10.1001/jama.2010.655. No abstract available. PMID 20501929
- [Result] F O Kern E, Beischel S, Stalnaker R, Aron DC, Kirsh SR, Watts SA. Building a diabetes registry from the Veterans Health Administration's computerized patient record system. J Diabetes Sci Technol. 2008 Jan;2(1):7-14. doi: 10.1177/193229680800200103. PMID 19885172

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemedicine CBOC: Designated CBOC's were involved in the intervention phase where their DM patients were asked to participate in a telemedicine visit.
  The Diabetes Treatment Satisfaction Questionnaire: A six question likert scale questionnaire regarding the patients treatment satisfaction. The responses range from very dissatisfied to very satisfied.
  Diabetes Empowerment Scale: A twenty-eight question likert scale questionnaire regarding the patients attitude towards diabetes. The responses range from strongly agree to strongly disagree.
  CBOC's undergo half-day joint-clinics via teleconference: A patient has Diabetes/Endo clinic visit via teleconferencing. A patient is at a CBOC and the Diabetes/Endo physician is at Wade Park.
- Provider Interview: Qualitative interviews with providers
Period: Overall Study
Arm/Group | Telemedicine CBOC | Control CBOC | Provider Interview
Started | 199 | 83 | 22
Completed | 199 | 83 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cohort I will consist of high-risk patients referred to a specialist during the 9-month active intervention and enrollment phase.Cohort II will consist of all other patients with diabetes (i.e., all non-Cohort I patients). We didn't collect gender or the complete age data.
  Qualitative interviews with providers
Groups:
- Telemedicine CBOC: Designated CBOC's were involved in the intervention phase where their DM patients were asked to participate in a telemedicine visit.
  The Diabetes Treatment Satisfaction Questionnaire: A six question likert scale questionnaire regarding the patients treatment satisfaction. The responses range from very dissatisfied to very satisfied.
  Diabetes Empowerment Scale: A twenty-eight question likert scale questionnaire regarding the patients attitude towards diabetes. The responses range from strongly agree to strongly disagree.
  CBOC's undergo half-day joint-clinics via teleconference: A patient has Diabetes/Endo clinic visit via teleconferencing. A patient is at a CBOC and the Diabetes/Endo physician is at Wade Park.
  We did not collect gender and age related data.
- Total: Total of all reporting groups
Arm/Group | Telemedicine CBOC | Control CBOC | Provider Interview | Total
Number analyzed (Participants) | 199 | 83 | 22 | 304
Age, Customized [Number; unit: participants]
  18 years and older | 199 | 83 | 22 | 304
Sex/Gender, Customized [Number; unit: participants] | NA — Gender was not collected for this study | NA — Gender was not collected for this study | NA — Gender was not collected for this study | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Secondary Outcome: Patient Satisfaction
Description: Diabetes Treatment Satisfaction Questionnaire (DTSQ) consists of 6 questions and ranges from 0-6. The following aspects of current treatment included were convenience, flexibility, understanding and continuing present form of treatment. The total range of the DTSQ is the sum of the 6 individual questions scores (i.e. 0-36) Higher scores represent greater satisfaction/convenience.
Time Frame: Base line and at18 months.
Population: The number subjects was determined on the size of the CBOC.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Telemedicine CBOC: Designated CBOC's were involved in the intervention phase where their DM patients were asked to participate in a telemedicine visit.
  The Behavioral: The Diabetes Treatment Satisfaction Questionnaire given during this phase along with the Behavioral: Diabetes Empowerment Scale and the Behavioral: CBOC's undergo half-day joint-clinics via teleconference.
  The Diabetes Treatment Satisfaction Questionnaire: A six question likert scale questionnaire regarding the patients treatment satisfaction. The responses range from very dissatisfied to very satisfied.
  Diabetes Empowerment Scale: A twenty-eight question likert scale questionnaire regarding the patients attitude towards diabetes. The responses range from strongly agree to strongly disagree.
  CBOC's undergo half-day joint-clinics via teleconference: A patient has Diabetes/Endo clinic visit via teleconferencing. A patient is at a CBOC and the Diabetes/Endo physician is at Wade Park.
- Control CBOC: Received the questionnaires by mail and had no intervention of diabetes teleconference
Arm/Group | Telemedicine CBOC | Control CBOC
Number analyzed (Participants) | 199 | 83
units on a scale
  baseline | 24.33 [0 to 36] | 23.29 [6 to 36]
  18 months | 23.55 [8 to 36] | 23.9 [8 to 36]
Statistical Analysis 1: Comparison: Telemedicine CBOC vs Control CBOC; Comparisons were made between the intervention and control groups at baseline; Test type: Superiority or Other; p > 0.153, t-test, 2 sided — Threshold for statistical significance was p<0.025 using Bonferroni correction for 2 statistical tests
Statistical Analysis 2: Comparison: Telemedicine CBOC vs Control CBOC; Comparisons were made between the intervention and control groups at 18 months; Test type: Superiority or Other; p > 0.25, t-test, 2 sided — Threshold for statistical significance was p<0.025 using Bonferroni correction for 2 statistical tests; Threshold for statistical significance was p<0.025 using Bonferroni correction for 2 statistical tests

2. Primary Outcome: A1c
Description: Hemoglobin A1c is a measure of glycemic control
Time Frame: baseline and 18 months
Measure: Mean (Full Range); unit: percentage of Hb that is glycosylated
Groups:
- Telemedicine: Intervention group
- Control: non intervention group
Arm/Group | Telemedicine | Control
Number analyzed (Participants) | 199 | 83
percentage of Hb that is glycosylated
  baseline | 10.1 [6.4 to 14.9] | 9.32 [5.3 to 15.9]
  18 months | 8.82 [5 to 14] | 8.36 [6 to 13]

ADVERSE EVENTS:
Arm/Group | Telemedicine CBOC | Control CBOC | Provider Interviews
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/83 | 0/22
Other Adverse Events (participants affected / at risk) | 0/199 | 0/83 | 0/22

LIMITATIONS AND CAVEATS:
A potential factor jeopardizing both internal and external validity relates to fact that the consultation process may be very dependent on the particular individuals involved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No